CLINICAL TRIAL: NCT05996809
Title: Post-Market Clinical Follow-up Study for COSEAL® in Gynecologic Surgery
Brief Title: PMCF Study for COSEAL® in Gynecologic Surgery
Status: Completed | Type: Observational
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: BXU571781
Record Dates: First submitted 2023-08-11; First posted 2023-08-18 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Adhesion
Keywords: gynecological surgery, adhesion related morbidities
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients who underwent an index gynecologic surgery: The population will consist of patients who underwent an index gynecologic surgery (performed at least 2 years prior to the start of the study) during which COSEAL was used
  Interventions: Device: Coseal

INTERVENTIONS:
Device: Coseal — Adhesion reduction

SUMMARY:
The study is a single-arm, retrospective, chart review with a patient questionnaire intended to supplement the patient chart, when necessary. The population will consist of patients who underwent an index gynecologic surgery (performed at least 2 years prior to the start of the study) during which COSEAL was used as an adjunct to good surgical technique to reduce the incidence, severity, and extent of post-surgical adhesion formation. The purpose of the study is to detect the incidence of adhesion-related morbidities as measured by the proportion of adhesion-related readmissions, including reoperations in these patients.

Patient charts will be reviewed to collect the data on readmissions related to adhesions, If the patient chart has no record of adhesion related readmission within approximately 2 years of the index surgery, then a patient questionnaire will be sent. A questionnaire may still be sent if a patient chart has a record of adhesion related readmission within approximately 2 years of the index surgery and further clarification is needed. The questionnaire will collect information regarding readmission or reoperation directly or possibly related to adhesions following the index gynecologic surgical procedure at a hospital or outpatient clinic other than that of the index surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adult female patients who, at the time of surgery, were ≥18 years of age and who have undergone an index gynecologic surgery at least 2 years prior to the start of the study.
2. Patients in whom COSEAL was used for the reduction of post-surgical adhesion formation

Exclusion Criteria:

1. Patients who had frank infection in the abdominopelvic cavity at the time of the surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Data will be collected from adult female patient charts in whom COSEAL was used as an adjunct to good surgical technique to reduce the incidence, severity, and extent of post-surgical adhesion formation. Data will also be collected from the questionnaire responses, when necessary
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-05-08 (Actual)

PRIMARY OUTCOMES:
Incidence of hospital readmissions directly or possibly related to adhesions following the use of COSEAL in gynecologic surgery, approximately 2 years from the date of index surgery. | within 2 years of surgery
  Patient charts will be reviewed to collect the data on readmissions related to adhesions, which are defined as:
  * Directly related to adhesions (adhesiolysis, non-operative readmissions for adhesions, and adhesiolysis operations on female reproductive tract);
  * Possibly related to adhesions (gynecologic operations, abdominal surgery, and nonoperative readmissions);
  * Open or laparoscopic reoperations that could potentially be complicated by present adhesions

CONTACTS AND LOCATIONS:
Locations (2):
- Feinberg School of Medicine, Chicago, Illinois, United States
- Universita Campus Bio Medico di Roma, Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: Yes
Sharing of Clinical Trial Data: Baxter is committed to sharing clinical trial data with external medical experts and scientific researchers in the interest of advancing public health. As such, Baxter will supply anonymized Individual Patient Datasets (IPD) and supporting documents (synopsis of clinical study reports, protocol and SAP's)
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Upon approval of a legitimate research request.
Access Criteria: Research requests will be reviewed by qualified medical and scientific experts within the company. If Baxter agrees to the release of clinical data for research purposes, the requestor will be required to sign a data sharing agreement (DSA) in order to ensure protection of patient confidentiality and any intellectual property rights of Baxter prior to the release of any data.
URL: http://www.baxter.com/clinical-trial-transparency-and-data-sharing-policy